CLINICAL TRIAL: NCT04737018
Title: Impact of a Focal Muscle Vibration Protocol in Front of the the Anterior Tibial Muscle in the Subacute Post-stroke Period on Motor Recovery in Hemiplegic Patients.
Acronym: VIBRATAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20CH152; 2020-A03189-30 (Other: ANSM)
Record Dates: First submitted 2021-01-28; First posted 2021-02-03 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: muscle vibration protocol; anterior tibia muscle; hemiplegic patient
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vibration program (Experimental): a 4-week program of muscular focal vibrations, at the rate of 5 sessions of 30 minutes per week, in addition to conventional rehabilitation. The program will apply a frequency of 100 Hz, with an amplitude of 1 mm
  Interventions: Other: Fugl-Meyer Assessment (FMA); Other: Medical Research Concil (MRC); Other: 2 Minute Walk Test (2MWT); Other: Timed Up & Go Test; Other: Modified Ashworth Scale; Other: Postural Assessment Scale for Stroke; Device: posturographic recording; Other: vibration program
- sham program (Sham Comparator): a 4-week program of muscular focal vibrations, at the rate of 5 sessions of 30 minutes per week, in addition to conventional rehabilitation.
  Interventions: Other: Fugl-Meyer Assessment (FMA); Other: Medical Research Concil (MRC); Other: 2 Minute Walk Test (2MWT); Other: Timed Up & Go Test; Other: Modified Ashworth Scale; Other: Postural Assessment Scale for Stroke; Device: posturographic recording; Other: sham program

INTERVENTIONS:
Other: Fugl-Meyer Assessment (FMA) — assessment of motor skills : measurement of the intensity of reflexes, as well as an assessment of voluntary movements and motor coordination Score from 0 to 34
Other: Medical Research Concil (MRC) — evaluation of muscular strength score from 0 to 5
Other: 2 Minute Walk Test (2MWT) — Assess functional walking and aerobic abilities
Other: Timed Up & Go Test — measures the time it takes to get up from a chair, walk 10 feet, turn around, return to the seat and sit down
Other: Modified Ashworth Scale — score from 0 to 4 evaluation of spasticity
Other: Postural Assessment Scale for Stroke — score from 0 to 36 measures the patient's ability to maintain stable postures and balance in changes of position
Device: posturographic recording — analysis of static equilibrium parameters and positional measurement of the center of gravity on the Winposturo platform
Other: vibration program — a 4-week program of muscular focal vibrations, at the rate of 5 sessions of 30 minutes per week, in addition to conventional rehabilitation. The program will apply a frequency of 100 Hz, with an amplitude of 1 mm
  Arms: vibration program
Other: sham program — a 4-week program of muscular focal vibrations, at the rate of 5 sessions of 30 minutes per week, in addition to conventional rehabilitation.
  Arms: sham program

SUMMARY:
In about 40 percent of cases, after a stroke, neuromotor impairment leads to activity limitations and the development of chronic functional disorders, which have a significant impact on patient autonomy.

In the early subacute phase, motor deficit in foot lifters is one of the factors limiting standing posture and ambulation, which is ultimately difficult to rehabilitate due to the lack of available techniques for obtaining early onset of useful active voluntary contraction.

The use of muscular focal vibration therapy, applied to relaxed muscle, may be of interest due to the portability and availability of the system and the neuromotor benefits demonstrated in healthy subjects and in acute and chronic post-stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Having had a stroke (with or without previous stroke) and being in the early subacute phase (between 14 days and 3 months of stroke).
* Responsible for a motor deficit in the right or left lower limb.
* No neurological history other than stroke.

Exclusion Criteria:

* Multifocal stroke
* Patient having received a botulinum toxin injection to the lower limb to be vibrated

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
score of Fugl Meyer Assessment (lower limbs) | day 30
  score from 0 to 34 Stroke-specific performance-based disability index that quantitatively assesses analytical motor skills in the lower limb.

SECONDARY OUTCOMES:
score of Fugl Meyer Assessment (lower limbs) | day 0, day 15, day 30 and month 2
  score from 0 to 34 Stroke-specific performance-based disability index that quantitatively assesses analytical motor skills in the lower limb.
score of Medical Research Concil | day 0, day 15, day 30 and month 2
  score of 0 (absence of contraction) to 5 (normal force)
assess functional walking ability | day 0, day 15, day 30 and month 2
  measured with 2 Minute Walk Test
score of postural assessment scale for stroke | day 0, day 15, day 30 and month 2
  measures the patient's ability to maintain stable postures, as well as balance in changes of position score of 0 (cannot perform the activity) to 36 (can perform the activity)
analysis of static equilibrium | day 0, day 15, day 30 and month 2
  with Winposturo platform
positional measurement of the center of gravity | day 0, day 15, day 30 and month 2
  with Winposturo platform

CONTACTS AND LOCATIONS:
Overall Officials: Bruno FERNANDEZ, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Saint-Etienne, Saint-Etienne
  - Le Clos Champirol - Service de Médecine Physique et de Réadaptation, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No